CLINICAL TRIAL: NCT01964651
Title: A Double-Blind, Placebo-Controlled, Randomized, Multiple Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of JNJ-42165279 in Healthy Young and Elderly Subjects
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of JNJ-42165279 in Healthy Young and Elderly Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR102575; 42165279EDI1002 (Other: Janssen Research & Development, LLC); 2013-002309-67 (EudraCT Number)
Record Dates: First submitted 2013-10-14; First posted 2013-10-17 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Healthy
Keywords: Healthy; JNJ-42165279; Pharmacokinetics; Elderly; Young
MeSH Terms: interventions — JNJ-42165279

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Cohort A (Part 1) (Experimental): Healthy male participants, 18 to 55 years of age.
  Interventions: Drug: JNJ-42165279 50 mg; Drug: Placebo
- Cohort B (Part 1) (Experimental): Healthy male participants, 18 to 55 years of age.
  Interventions: Drug: JNJ-42165279 30 mg; Drug: Placebo
- Cohort C (Part 2) (Experimental): Healthy female participants of nonchildbearing potential (surgically sterile or postmenopausal), 18 to 58 years of age.
  Interventions: Drug: JNJ-42165279 100 mg; Drug: Placebo
- Cohort D (Part 2) (Experimental): Healthy elderly male or female participants, from 65 to 85 years of age.
  Interventions: Drug: JNJ-42165279 100 mg; Drug: Placebo

INTERVENTIONS:
Drug: JNJ-42165279 50 mg — JNJ-42165279 50 mg orally administered once daily for 10 days.
  Arms: Cohort A (Part 1)
Drug: JNJ-42165279 100 mg — JNJ-42165279 100 mg orally administered once daily for 10 days.
  Arms: Cohort C (Part 2); Cohort D (Part 2)
Drug: JNJ-42165279 30 mg — JNJ-42165279 30 mg orally administered once daily for 10 days.
  Arms: Cohort B (Part 1)
Drug: Placebo — Matching placebo orally administered once daily for 10 days.

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and pharmacokinetics of JNJ-42165279 in healthy, young and elderly, male and female participants after repeated oral dose administration.

DETAILED DESCRIPTION:
This is a double-blind (neither physician nor participant knows the treatment that the participant receives), randomized (the study drug is assigned by chance), placebo-controlled (an inactive substance is compared with a medication to test whether the medication has a real effect in a clinical study) trial that will be conducted in two parts. Thirty two (32) healthy participants are planned to be included in total, in four cohorts (groups). Participants in each cohort will receive JNJ-42165279 (n=6) or placebo (n=2) once-daily for 10 consecutive days. In Part 1, two cohorts of healthy male participants, 18 to 55 years of age, will be enrolled. Cohort A will receive 50 mg JNJ-42165279 or placebo for 10 days, and Cohort B will receive 30 mg JNJ-42165279 or placebo for 10 days. In Part 2, Cohort C will consist of 8 healthy female participants of non-childbearing potential (surgically sterile or postmenopausal), 18 to 58 years of age, who will receive 100 mg JNJ-42165279 or placebo for 10 days. Cohort D will consist of 8 healthy elderly male or female participants, from 65 to 85 years of age, who will receive 100 mg JNJ-42165279 or placebo for 10 days. The dose may be adapted before each cohort starts based on available data. The maximum dose will not exceed 100 mg once-daily. For all participants, this study will consist of an eligibility screening examination (between 28 and 3 days prior to the first dose administration), a double-blind treatment phase consisting of 2 days before dosing, 10 dosing days (Day 1 to 10), 4 days after dosing (Day 11 to 14), and a follow-up examination (within 7 to 14 days after last dose administration). The total study duration for each participant will not exceed 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) between 18 and 30 kg/m2 inclusive
* Nonsmoker
* Healthy men between 18 and 55 years, inclusive (Cohorts A and B)
* Healthy women between 18 and 58 years, inclusive (Cohort C)
* Healthy men and women between 65 and 85 years of age, inclusive (Cohort D)
* Men who are sexually active with a woman of childbearing potential and have not had a vasectomy must agree to use a barrier method of birth control during the study and for 3 months after receiving the last dose of study drug. In addition, their female partners should also use an appropriate method of birth control for at least the same duration (Cohorts A, B, and D)
* Not be of childbearing potential due to either tubal ligation or hysterectomy, or who are postmenopausal (Cohorts C and D)

Exclusion Criteria:

* Clinically significant abnormal values for hematology, clinical chemistry or urinalysis at screening or admission
* Clinically significant abnormal physical examination, vital signs or electrocardiogram at screening or admission
* History of, or current, significant medical illness including (but not limited to) cardiac disease, hematological disease, lipid abnormalities, respiratory disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, Parkinson's disease, infection, or any other illness that the Investigator considers should exclude the participant
* History of epilepsy or fits or unexplained black-outs
* Cohorts A and B only: a contraindication for spinal puncture

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of JNJ-42165279 | 2 weeks
Urine concentrations of JNJ-42165279 | 2 weeks
Concentrations in cerebrospinal fluid of JNJ-42165279 | 2 weeks
The number of participants with adserve events as a measure of safety and tolerability | Approximately 8 weeks

SECONDARY OUTCOMES:
Enzyme fatty acid amide hydrolase inhibition, as measured in white blood cells (WBCs) | Approximately 4 weeks
Plasma concentrations of N-arachidonoylethanolamine (anandamide) | 2 weeks
Plasma concentrations of palmitoylethanolamide | 2 weeks
Plasma concentrations of oleoylethanolamide | 2 weeks
Serum concentrations of prolactin | 10 days
Saliva concentrations of cortisol | 10 days
Concentrations in cerebrospinal fluid of N-arachidonoylethanolamine (anandamide) or its metabolites | 9 days
Concentrations in cerebrospinal fluid of palmitoylethanolamide or its metabolites | 9 days
Concentrations in cerebrospinal fluid of oleoylethanolamide or its metabolites | 9 days

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Merksem, Belgium